CLINICAL TRIAL: NCT01184170
Title: Metabolically Normal and Metabolically Abnormal Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10-0708
Record Dates: First submitted 2010-08-12; First posted 2010-08-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: obesity; metabolism; cardiovascular metabolic syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metabolically Normal (Experimental): Subjects in this group are metabolically normal. They have low liver fat defined as less than five percent as determined by magnetic resonance spectroscopy.
  Intervention: Subjects will begin an 8-12 week high-calorie diet intervention. They will eat an additional 1000 kcal/day for two to three months, until a moderate, approximately 5% weight gain is achieved. The recommended dietary energy intake will be 1000 kcal/d more than the subject's baseline resting energy expenditure. An individualized diet plan will be developed for each subject by the study dietitian based on estimated energy requirements, and the subject's food preferences and dietary habits.
  Interventions: Behavioral: overfeeding
- Metabolically Abnormal (Experimental): Subjects in this group are metabolically abnormal. They have high liver fat defined as at least ten percent as determined by magnetic resonance spectroscopy.
  Intervention: Subjects will begin an 8-12 week high-calorie diet intervention. They will eat an additional 1000 kcal/day for two to three months, until a moderate, approximately 5% weight gain is achieved. The recommended dietary energy intake will be 1000 kcal/d more than the subject's baseline resting energy expenditure. An individualized diet plan will be developed for each subject by the study dietitian based on estimated energy requirements, and the subject's food preferences and dietary habits.
  Interventions: Behavioral: overfeeding

INTERVENTIONS:
Behavioral: overfeeding — Subjects will begin an 8-12 week high-calorie diet intervention. They will eat an additional 1000 kcal/day for two to three months, until a moderate, approximately 5% weight gain is achieved. The recommended dietary energy intake will be 1000 kcal/d more than the subject's baseline resting energy expenditure. An individualized diet plan will be developed for each subject by the study dietitian based on estimated energy requirements, and the subject's food preferences and dietary habits.
  Other Names: directed weight gain

SUMMARY:
The purpose of this study is to learn more about why some obese persons are resistant to developing obesity-related metabolic diseases (such as diabetes and cardiovascular disease), while others are prone to developing these conditions. We will do this by studying obese persons before and after a 5% body weight gain.

Subjects will be asked to increase their current diet for a period of 8-12 weeks in order to increase their current body weight by 5%. Each will then be asked to maintain this weight increase for 3 weeks. We will monitor subjects throughout this time period with weekly medical evaluations. At the completion of the study, we will provide each subject with a 6-month weight loss program.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects (BMI 30.0 - 39.9 kg/m2)
* Sedentary subjects (exercise less than 1 hr/wk)

Exclusion Criteria:

* Pregnant or lactating women
* Michigan Alcohol Screening Test score ≥4
* Active or previous history of liver disease
* Active or previous history of diabetes
* history of alcohol abuse, or currently consuming ≥20 g alcohol/day
* Severe hypertriglyceridemia (>300 mg/dL)
* Smoke tobacco
* Take medication that might confound the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in Intrahepatic Triglyceride | an average of three months, from baseline to 5% weight gain
Change in de novo lipogenesis | an average of three months, from baseline to 5% weight gain
Change in VLDL kinetics | an average of three months, from baseline to 5% weight gain
Change in hepatic insulin sensitivity | an average of three months, from baseline to 5% weight gain
Change in skeletal muscle insulin sensitivity | an average of three months, from baseline to 5% weight gain

SECONDARY OUTCOMES:
Change in adipose tissue insulin sensitivity | an average of three months, from baseline to 5% weight gain
Change in CD36 concentration in skeletal muscle | an average of three months, from baseline to 5% weight gain
change in CD36 concentration in adipose tissue | an average of three months, from baseline to 5% weight gain
Change in cell proliferation (growth) rates in the colon | an average of three months, from baseline to 5% weight gain

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Yoshino J, Patterson BW, Klein S. Adipose Tissue CTGF Expression is Associated with Adiposity and Insulin Resistance in Humans. Obesity (Silver Spring). 2019 Jun;27(6):957-962. doi: 10.1002/oby.22463. Epub 2019 Apr 19. PMID 31004409
- [Derived] Fabbrini E, Tiemann Luecking C, Love-Gregory L, Okunade AL, Yoshino M, Fraterrigo G, Patterson BW, Klein S. Physiological Mechanisms of Weight Gain-Induced Steatosis in People With Obesity. Gastroenterology. 2016 Jan;150(1):79-81.e2. doi: 10.1053/j.gastro.2015.09.003. Epub 2015 Sep 12. PMID 26376348
- [Derived] Fabbrini E, Yoshino J, Yoshino M, Magkos F, Tiemann Luecking C, Samovski D, Fraterrigo G, Okunade AL, Patterson BW, Klein S. Metabolically normal obese people are protected from adverse effects following weight gain. J Clin Invest. 2015 Feb;125(2):787-95. doi: 10.1172/JCI78425. Epub 2015 Jan 2. PMID 25555214